CLINICAL TRIAL: NCT06026787
Title: Clinical Value of Adding Dapagliflozin in Patients With Nephrotic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS 419/2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Nephrotic Syndrome; Sodium-Glucose Transporter 2 Inhibitors
MeSH Terms: conditions — Nephrotic Syndrome | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin Arm (Experimental): During the study duration of 6 months, this cohort will be administered a daily dose of 10 mg dapagliflozin in conjunction with the standard of care for primary nephrotic syndrome based on the KDIGO 2021 guidelines. The conventional treatment regimen may encompass immunosuppressive medications, agents that block the renin-angiotensin-aldosterone system (RAAS), statins, and diuretics as deemed necessary.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control Arm (No Intervention): This cohort will exclusively be subjected to the standard of care tailored for primary nephrotic syndrome. This could encompass administration of immunosuppressive drugs, agents targeting the renin-angiotensin-aldosterone system (RAAS), statins, and diuretics as warranted by individual needs.

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg will be added to the standard of care regimen of primary nephrotic syndrome patients
  Arms: Dapagliflozin Arm

SUMMARY:
Conducted as a randomized controlled clinical trial, this study aims to assess the potential benefits of incorporating dapagliflozin, an SGLT-2 inhibitor, into the treatment regimen of patients diagnosed with primary nephrotic syndrome. The primary focus is on examining the impact of dapagliflozin on two key parameters: proteinuria and estimated glomerular filtration rate (eGFR).

The trial involves adult participants who have been definitively diagnosed with primary nephrotic syndrome through renal biopsy. In conjunction with their standard care, these participants will receive a daily dose of dapagliflozin at 10 mg. Over a span of six months, they will undergo comprehensive monthly assessments. These assessments will involve the collection and analysis of urine samples to quantify proteinuria and perform urinalysis. Additionally, blood samples will be taken to determine the estimated eGFR, lipid profile, glycated hemoglobin. Participants will also be encouraged to report any potential side effects resulting from their medication intake.

ELIGIBILITY:
Inclusion Criteria:

* eGFR > 25 mL/min/1.73m2
* Evidence of primary nephrotic syndrome by renal biopsy
* Non-diabetic kidney disease

Exclusion Criteria:

* Nephrotic syndrome secondary to lupus nephritis, AAV, amyloidosis, or secondary membranous nephropathy
* Hepatic impairment [AST or ALT >3 times ULN or total bilirubin >2 times the ULN] at the time of enrolment
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Proteinuria | 6 months
  Effect of dapagliflozin on proteinuria
Estimated GFR | 6 months

OTHER OUTCOMES:
Lipid profile | 6 months
Body Weight | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt